CLINICAL TRIAL: NCT01490333
Title: Sunweavers: Supporting Native American Women's Vitamin D Research
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: H-2010-0118
Record Dates: First submitted 2011-11-29; First posted 2011-12-12 (Estimated); Last update posted 2014-11-20 (Estimated); Status verified 2014-11

CONDITIONS: Vitamin D Deficiency; Cardiovascular Diseases
MeSH Terms: conditions — Vitamin D Deficiency; Cardiovascular Diseases | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2500 IU Vitamin D3 (Experimental)
  Interventions: Dietary Supplement: Vitamin D3
- 400 IU Vitamin D3 (Active Comparator)
  Interventions: Dietary Supplement: Vitamin D3

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — The vitamin D3 will be taken daily.

SUMMARY:
Cardiovascular disease (CVD) and diabetes occur commonly among Native Americans (NA), and are leading causes of death among northern US NAs. Moreover, low vitamin D status occurs commonly in this same population. An increasing amount of evidence indicates a correlation between low vitamin D status and CVD and diabetes by contributing to a heightened pro-inflammatory environment within the endothelial lining of blood vessels leading to atherosclerotic disease, and an impaired sensitivity to insulin leading to diabetes. Our fundamental hypothesis is that low vitamin D status is a risk factor for CVD by causing a proinflammatory milieu, thereby leading to endothelial dysfunction. Additionally, the investigators hypothesize that vitamin D supplementation will reduce inflammation, thereby restoring endothelial function and ultimately reducing CVD risk.

DETAILED DESCRIPTION:
Low vitamin D status is endemic due to 21st century lifestyle, which limits sun exposure, and inadequate dietary intake. An increasing body of data relates low vitamin D status to increased risk for non-musculoskeletal morbidities including, most notably, cardiovascular disease (CVD) and type II diabetes mellitus (T2DM). CVD, for which T2DM is a major risk factor, causes over one-third of all deaths in the US. Moreover, American Indians (AI) and Alaskan Natives (AN) are 20% more likely to develop CVD and 2.2 times more likely to develop DM than non-Hispanic whites. In fact, AI of the Great Lakes Region (Bemidji Area) have the third highest DM rate in the nation, an age-adjusted DM mortality rate almost three-fold higher than the all-race mortality, and the highest rates of CVD among AI nationally. In this population, where CVD and DM are two of the top four causes of death, our preliminary work finds low vitamin D status commonplace.

As low vitamin D status, CVD and T2DM are epidemic among AI, the investigators hypothesize that low vitamin D is causally related to CVD and T2DM by establishing a pro-inflammatory milieu, which in turn predisposes to CVD and T2DM. As such, vitamin D supplementation should reduce markers of inflammation and thereby ultimately reduce risk for CVD and T2DM. This work will explore this possibility by evaluating the effect of vitamin D status on endothelial function (measured by arterial reactivity), plasma biomarkers of inflammation and glucose homeostasis in 100 postmenopausal AI women. Subjects will receive vitamin D3, either 400 or 2,500 IU, daily for six months. The investigators will define the effects of vitamin D status, and subsequent response to supplementation, on endothelial function, arterial stiffness (flow-mediated vasodilation (FMD) of the brachial artery, and carotid to femoral pulse wave velocity (PWV)), plasma markers of inflammation and glucose homeostasis. All study participants will have fasting laboratory and noninvasive vascular ultrasound studies performed at baseline and following three and six months of study. Plasma concentration of pro-inflammatory cytokines will be measured as secondary outcome variables. Fasting blood glucose, insulin and the adipocytokines leptin and adiponectin, will be measured as exploratory outcomes for potential future studies.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory, community dwelling AI woman
* Postmenopausal up to age 75 years; for women below age 55, postmenopausal status must be confirmed by documentation of serum FSH>30 IU/L and estradiol < 20 pg/ml unless a bilateral oophorectomy is documented.

Exclusion Criteria:

* Serum 25(OH)D < 10 or > 60 ng/ml.
* Known CVD (history of MI, coronary artery bypass graft surgery, percutaneous coronary intervention, stroke, transient ischemic attack, peripheral arterial disease with claudication).
* Uncontrolled thyroid disease (thyroid stimulating hormone level outside of normal range).
* Change in dose of lipid lowering medications within the preceding six weeks.
* Mastectomy of the right breast
* Non-English speaking, illiterate, impaired decision making.

Ages: 55 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2011-07; Primary Completion 2014-01 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Change in markers of endothelial function | Baseline visit, 3 month visit and 6 month visit.
  This will be determined by evaluating CRP and lipid panel
Change in arterial stiffness with vitamin D3 supplementation | one year
  Change in arterial stiffness will be evaluated with radial tonometry.

SECONDARY OUTCOMES:
Plasma concentration of pro-inflammatory cytokines | Baseline visit, 3 month visit, and 6 month visit.
  This will be evaluated by assessing TNF alpha, IL6, VCAM and ICAM

CONTACTS AND LOCATIONS:
Overall Officials: Neil Binkley, M.D., Principal Investigator — University of Wisconsin, Madison
Locations (3):
- United States (3):
  - Stockbridge-Munsee Nation, Bowler, Wisconsin
  - Bad River Nation, Lac du Flambeau, Wisconsin
  - University of Wisconsin Osteoporosis Clinical Research Program, Madison, Wisconsin

REFERENCES:
- [Derived] Gepner AD, Haller IV, Krueger DC, Korcarz CE, Binkley N, Stein JH. A randomized controlled trial of the effects of vitamin D supplementation on arterial stiffness and aortic blood pressure in Native American women. Atherosclerosis. 2015 Jun;240(2):526-8. doi: 10.1016/j.atherosclerosis.2015.04.795. Epub 2015 Apr 25. PMID 25955191